CLINICAL TRIAL: NCT00508261
Title: Co-Administration of GSK Biologicals' Meningococcal Vaccine GSK134612 With Infanrix Hexa™, Compared to Individual Administration of Each Vaccine, in Healthy 12- Through 23-Month-Old Children
Brief Title: Co-Administration of Meningococcal Vaccine GSK134612 With Infanrix Hexa™ Versus Individual Administration of Each Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109835
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2017-05

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal vaccine; Immunogenicity; Routine infancy vaccination; Safety
MeSH Terms: conditions — Meningococcal Infections

ARMS (4):
- Group A (Experimental): Meningococcal vaccine GSK134612 co-administered with Infanrix hexa™
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Infanrix™ hexa
- Group B (Experimental): Meningococcal vaccine GSK134612 followed one month later by Infanrix hexa™
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Infanrix™ hexa
- Group C (Active Comparator): Infanrix hexa™ followed one month later by Meningococcal vaccine GSK134612
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Infanrix™ hexa
- Group D (Active Comparator): Meningitec™ vaccination
  Interventions: Biological: Meningitec™

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — Single dose intramuscular injection
  Arms: Group A; Group B; Group C
Biological: Infanrix™ hexa — Single dose intramuscular injection
  Arms: Group A; Group B; Group C
Biological: Meningitec™ — Single dose intramuscular injection
  Arms: Group D

SUMMARY:
The purpose of this study is to demonstrate, in 12-23 months old subjects, the non-inferiority of meningococcal vaccine GSK134612 co-administered with Infanrix hexa™, compared to each vaccine administered individually and to licensed meningococcal vaccine Meningitec™.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Multicentre study with 4 parallel groups. One group will receive GSK134612 co-administered with Infanrix hexa™, two groups will receive sequential administration of GSK134612 and Infanrix hexa™ and the final group will receive Meningitec™.

For subjects in Groups B and C, three blood samples will be taken: prior to first vaccination and 1 month after each vaccination.

For subjects in Groups A and D, two blood samples will be taken: prior to and 1 month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 23 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Documented three-dose primary vaccination with DTPa, hepatitis B, inactivated polio and Haemophilus influenzae type b conjugate vaccines, completed at least 180 days before administration of the first study vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of any vaccine not foreseen by the study protocol, including measles, mumps, rubella, varicella and pneumococcal vaccines, within 30 days before the first dose of vaccine(s) and 30 days after the last dose of vaccine(s).
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W and/or Y.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C, W and/or Y.
* Previous booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis or Haemophilus influenzae type b.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Additional criteria for subjects receiving Infanrix hexa™

* Hypersensitivity reaction due to previous vaccination with Infanrix hexa™.
* Encephalopathy defined as an acute, severe central nervous system disorder occurring within 7 days following vaccination and generally consisting of major alterations in consciousness, unresponsiveness, generalised or focal seizures that persist more than a few hours, with failure to recover within 24 hours.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 793 (Actual)
Dates: Start 2007-08-01; Primary Completion 2008-05-26 (Actual); Study Completion 2008-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (76):
- Austria (5):
  - GSK Investigational Site, Eferding
  - GSK Investigational Site, Neufeld/Leitha
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Villach
  - GSK Investigational Site, Wels
- Germany (65):
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Heilbronn, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Marbach, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Pforzheim, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Kaufbeuren, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Kronach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Braunatal, Hesse
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wildeshausen, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Balve, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Datteln, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Espelkamp, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gau-Odernheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Oppenheim, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Stollberg, Saxony
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Didimoteicho
  - GSK Investigational Site, Karditsa
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Véria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Knuf M, Pantazi-Chatzikonstantinou A, Pfletschinger U, Tichmann-Schumann I, Maurer H, Maurer L, Fischbach T, Zinke H, Pankow-Culot H, Papaevangelou V, Bianco V, Van der Wielen M, Miller JM. An investigational tetravalent meningococcal serogroups A, C, W-135 and Y-tetanus toxoid conjugate vaccine co-administered with Infanrix hexa is immunogenic, with an acceptable safety profile in 12-23-month-old children. Vaccine. 2011 Jun 6;29(25):4264-73. doi: 10.1016/j.vaccine.2011.03.009. Epub 2011 Mar 21. PMID 21420417
- [Background] Maurer H et al. Co-administration of MENACWY-TT conjugate vaccine with DTPA-HBV-IPV/HIB vaccine does not impair immune response to DTPA-HBV-IPV/HIB, and has an acceptable safety profile. Abstract presented at the 28th Annual Meeting of European Society for Paediatric Infectious Diseases (ESPID). Nice, France, 4-8 May 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109835 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix + Infanrix-hexa Group: Subjects received concomitant administration of 1 dose of Nimenrix™ and Infanrix-hexa™ vaccines at Day 0.
- Nimenrix Group: Subjects received a single dose of Nimenrix™ vaccine at Day 0, followed one month later by 1 dose of Infanrix-hexa™ vaccine.
- Infanrix-Hexa Group: Subjects received a single dose of Infanrix-Hexa™ vaccine at Day 0, followed one month later by 1 dose of Nimenrix™ vaccine.
- Meningitec Group: Subjects received 1 dose of Meningitec™ vaccine at Day 0 and were permitted to receive the routinely recommended Infanrix-hexa booster once the active safety follow-up of this study was completed.
Period: Overall Study
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Started | 222 | 220 | 224 | 127
Completed | 219 | 212 | 218 | 126
Not Completed | 3 | 8 | 6 | 1
Not completed — Other | 0 | 1 | 1 | 0
Not completed — Serious Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 4 | 0
Not completed — Migrated/ moved from study area | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group | Total
Number analyzed (Participants) | 222 | 220 | 224 | 127 | 793
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.6 (3.01) | 15 (3.33) | 14.9 (3.17) | 14.6 (2.99) | 14.8 (3.14)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 109 | 106 | 119 | 61 | 395
  Male | 113 | 114 | 105 | 66 | 398
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian/ European heritage, n (%) | 204 | 205 | 212 | 120 | 741
  African heritage / African American | 3 | 4 | 1 | 2 | 10
  American Indian or Alaskan native | 2 | 1 | 0 | 1 | 4
  Asian - Central/ South Asian heritage | 1 | 2 | 1 | 0 | 4
  Asian - East Asian heritage | 2 | 0 | 0 | 0 | 2
  Asian - South east Asian heritage | 2 | 0 | 4 | 2 | 8
  White - Arabic / North African heritage | 4 | 7 | 4 | 2 | 17
  Other | 4 | 1 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers ≥ the Cut-off.
Description: The cut-off for the assay was greater than or equal to (≥) 1:8. The analysis was based only on subjects receiving Nimenrix vaccination at Day 0.
Time Frame: 1 month after vaccination with Nimenrix vaccine (Month 1)
Population: The analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group
Number analyzed (Participants) | 193 | 186
Participants
  rSBA-MenA, M1: number analyzed (Participants) | 193 | 183
  rSBA-MenA, M1 | 193 | 180
  rSBA-MenC, M1: number analyzed (Participants) | 191 | 183
  rSBA-MenC, M1 | 191 | 178
  rSBA-MenW-135, M1 | 193 | 183
  rSBA-MenY, M1: number analyzed (Participants) | 192 | 185
  rSBA-MenY, M1 | 192 | 180
Statistical Analysis 1: Comparison: Nimenrix + Infanrix-hexa Group vs Nimenrix Group; Demonstration of the non-inferiority of Nimenrix vaccine co-administered with combined Infanrix-hexa vaccine given alone in terms of bactericidal antibodies to Neisseria meningitidis serogroup A, at month 1; Test type: Non-Inferiority — Criterion for non-inferiority: The lower limit of the two-sided standardized asymptotic 95% confidence interval (CI) for the group difference in the percentages of subjects with serum bactericidal antibodies using baby rabbit complement (rSBA) titer ≥1:8 is greater than or equal to the pre-defined clinical limit of -10%; Difference in percentages = 1.64, 95% CI 2-sided [-0.33 to 4.71]
Statistical Analysis 2: Comparison: Nimenrix + Infanrix-hexa Group vs Nimenrix Group; Demonstration of the non-inferiority of the Nimenrix vaccine co-administered with combined Infanrix-hexa vaccine given alone in terms of bactericidal antibodies to Neisseria meningitidis serogroup C, at month 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 2.73, 95% CI 2-sided [0.73 to 6.24]
Statistical Analysis 3: Comparison: Nimenrix + Infanrix-hexa Group vs Nimenrix Group; Demonstration of the non-inferiority of the Nimenrix vaccine co-administered with combined Infanrix-hexa vaccine given alone in terms of bactericidal antibodies to Neisseria meningitidis serogroup W-135, at month 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 1.61, 95% CI 2-sided [-0.36 to 4.64]
Statistical Analysis 4: Comparison: Nimenrix + Infanrix-hexa Group vs Nimenrix Group; Demonstration of the non-inferiority of the Nimenrix vaccine co-administered with combined Infanrix-hexa vaccine given alone in terms of bactericidal antibodies to Neisseria meningitidis serogroup Y, at month 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 2.7, 95% CI 2-sided [0.71 to 6.18]

2. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Concentrations
Description: The analysis was based only on subjects receiving Infanrix-hexa vaccination. The results were calculated as geometric mean expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: 1 month after the first vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.The analysis for the primary outcome was based only on subjects receiving Infanrix-hexa vaccination at month 1.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Infanrix-Hexa Group
Number analyzed (Participants) | 191 | 179
EL.U/mL
  Anti-PT, M1 | 86 [77 to 95] | 85 [75 to 96]
  Anti-FHA, M1 | 542 [492 to 597] | 544 [485 to 611]
  Anti-PRN, M1 | 470 [411 to 537] | 450 [387 to 522]
Statistical Analysis 1: Comparison: Nimenrix + Infanrix-hexa Group vs Infanrix-Hexa Group; Demonstration of non-inferiority of combined Infanrix-hexa vaccine co-administered with Nimenrix vaccine to Infanrix-hexa vaccine given alone in terms of geometric mean concentrations (GMCs) of antibodies to pertussis toxoid (PT), at month 1; Test type: Non-Inferiority — Criterion for non-inferiority (1 month after the first study vaccination): The lower limit of the two-sided 95% CI on the GMC ratio for anti-PT (ELISA) is greater than or equal to a pre-defined clinical limit of delta = 0.67; Adjusted GMC ratios = 0.97, 95% CI 2-sided [0.83 to 1.12]
Statistical Analysis 2: Comparison: Nimenrix + Infanrix-hexa Group vs Infanrix-Hexa Group; Demonstration of non-inferiority of combined Infanrix-hexa vaccine co-administered with Nimenrix vaccine to Infanrix-hexa vaccine given alone in terms of geometric mean concentrations (GMCs) of antibodies to filamentous haemagglutinin (FHA), at month 1; Test type: Non-Inferiority — Criterion for non-inferiority (1 month after the first study vaccination): The lower limit of the two-sided 95% CI on the GMC ratio for anti-FHA (ELISA) is greater than or equal to a pre-defined clinical limit of delta = 0.67; Adjusted GMC ratios = 0.98, 95% CI 2-sided [0.85 to 1.13]
Statistical Analysis 3: Comparison: Nimenrix + Infanrix-hexa Group vs Infanrix-Hexa Group; Demonstration of non-inferiority of combined Infanrix-hexa vaccine co-administered with Nimenrix vaccine to Infanrix-hexa vaccine given alone in terms of geometric mean concentrations (GMCs) of antibodies to pertactin (PRN), at month 1; Test type: Non-Inferiority — Criterion for non-inferiority (1 month after the first study vaccination): The lower limit of the two-sided 95% CI on the GMC ratio for anti-PRN (ELISA) is greater than or equal to a pre-defined clinical limit of delta = 0.67; Adjusted GMC ratios = 0.92, 95% CI 2-sided [0.78 to 1.1]

3. Primary Outcome: Number of Subjects With Anti-HBs Concentrations ≥ the Cut-off
Description: The cut-off for the assay was greater than or equal to (≥) 10 milli-interantional units per milliliter (mIU/mL).
Time Frame: 1 month after vaccination with Nimenrix vaccine (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination. The analysis for the primary outcome measure was based only on subjects receiving Infanrix-hexa vaccination at Month 1.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix + Infanrix-hexa Group: Subjects received concomitant administration of 1 dose of Nimenrix and Infanrix-hexa vaccines at Day 0.
- Infanrix-Hexa Group: Subjects received a single dose of Infanrix-Hexa vaccine at Day 0, followed one month later by 1 dose of Nimenrix vaccine.
Arm/Group | Nimenrix + Infanrix-hexa Group | Infanrix-Hexa Group
Number analyzed (Participants) | 181 | 169
Participants | 180 | 166
Statistical Analysis 1: Comparison: Nimenrix + Infanrix-hexa Group vs Infanrix-Hexa Group; Test type: Non-Inferiority — Criterion for non-inferiority (1 month after the first study vaccination): The lower limit of the two-sided standardized asymptotic 95% CI for the group difference in the percentages of subjects with anti-HBs antibody concentrations ≥10 mIU/ml is greater than or equal to the pre-defined clinical limit of -10%; Difference in percentages = 1.22, 95% CI 2-sided [-1.47 to 4.6]

4. Primary Outcome: Number of Subjects With Anti-PRP Concentrations ≥ the Cut-off
Description: The cut-off for the assay was ≥ 1μg/mL.
Time Frame: 1 month after vaccination with Nimenrix vaccine (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.The analysis for the primary outcome was based only on subjects receiving Infanrix-hexa vaccination at Day 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Infanrix-Hexa Group
Number analyzed (Participants) | 184 | 173
Participants | 183 | 170
Statistical Analysis 1: Comparison: Nimenrix + Infanrix-hexa Group vs Infanrix-Hexa Group; Test type: Non-Inferiority — Criterion for non-inferiority (1 month after the first study vaccination): The lower limit of the two-sided standardized asymptotic 95% CI for the group difference in the percentage of subjects with anti-PRP concentrations (ELISA) ≥1.0 μg/mL is greater than or equal to the pre-defined clinical limit of -10%; Difference in percentages = 1.19, 95% CI 2-sided [-1.45 to 4.5]

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 1:8 and ≥ 1:128
Time Frame: At month 0, month 1 and month 2
Population: ATP cohort for immunogenicity, including all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination. Subjects in "Nimenrix + Infanrix-hexa Group" and "Meningitec Group" only had 2 blood samples taken: prior to (M0) and 1 month after vaccination (M1).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 193 | 186 | 179 | 114
Participants
  rSBA-MenA [M 0], ≥1:8: number analyzed (Participants) | 84 | 77 | 72 | 46
  rSBA-MenA [M 0], ≥1:8 | 30 | 32 | 34 | 18
  rSBA-MenA [M 1], ≥1:8: number analyzed (Participants) | 193 | 183 | 163 | 100
  rSBA-MenA [M 1], ≥1:8 | 193 | 180 | 71 | 43
  rSBA-MenA [M 2], ≥1:8: number analyzed (Participants) | 0 | 90 | 178 | 0
  rSBA-MenA [M 2], ≥1:8 |  | 90 | 178 |
  rSBA-MenA [M 0], ≥1:128: number analyzed (Participants) | 84 | 77 | 72 | 46
  rSBA-MenA [M 0], ≥1:128 | 18 | 21 | 24 | 11
  rSBA-MenA [M 1], ≥1:128: number analyzed (Participants) | 193 | 183 | 163 | 100
  rSBA-MenA [M 1], ≥1:128 | 193 | 179 | 57 | 30
  rSBA-MenA [M 2], ≥1:128: number analyzed (Participants) | 0 | 90 | 178 | 0
  rSBA-MenA [M 2], ≥1:128 |  | 90 | 178 |
  rSBA-MenC [M 0], ≥1:8: number analyzed (Participants) | 93 | 91 | 92 | 54
  rSBA-MenC [M 0], ≥1:8 | 20 | 25 | 13 | 11
  rSBA-MenC [M 1], ≥1:8: number analyzed (Participants) | 191 | 183 | 177 | 114
  rSBA-MenC [M 1], ≥1:8 | 191 | 178 | 34 | 112
  rSBA-MenC [M 2], ≥1:8: number analyzed (Participants) | 0 | 94 | 178 | 0
  rSBA-MenC [M 2], ≥1:8 |  | 91 | 178 |
  rSBA-MenC [M 0], ≥1:128: number analyzed (Participants) | 93 | 91 | 92 | 54
  rSBA-MenC [M 0], ≥1:128 | 5 | 8 | 5 | 3
  rSBA-MenC [M 1], ≥1:128: number analyzed (Participants) | 191 | 183 | 177 | 114
  rSBA-MenC [M 1], ≥1:128 | 189 | 172 | 14 | 102
  rSBA-MenC [M 2], ≥1:128: number analyzed (Participants) | 0 | 94 | 178 | 0
  rSBA-MenC [M 2], ≥1:128 |  | 85 | 157 |
  rSBA-MenW-135 [M 0], ≥1:8: number analyzed (Participants) | 91 | 84 | 85 | 55
  rSBA-MenW-135 [M 0], ≥1:8 | 43 | 42 | 46 | 22
  rSBA-MenW-135 [M 1], ≥1:8: number analyzed (Participants) | 193 | 186 | 173 | 112
  rSBA-MenW-135 [M 1], ≥1:8 | 193 | 183 | 86 | 41
  rSBA-MenW-135 [M 2], ≥1:8: number analyzed (Participants) | 0 | 91 | 179 | 0
  rSBA-MenW-135 [M 2], ≥1:8 |  | 91 | 179 |
  rSBA-MenW-135 [M 0], ≥1:128: number analyzed (Participants) | 91 | 84 | 85 | 55
  rSBA-MenW-135 [M 0], ≥1:128 | 17 | 11 | 23 | 10
  rSBA-MenW-135 [M 1] ≥1:128: number analyzed (Participants) | 193 | 186 | 173 | 112
  rSBA-MenW-135 [M 1] ≥1:128 | 193 | 180 | 49 | 23
  rSBA-MenW-135 [M 2], ≥1:128: number analyzed (Participants) | 0 | 91 | 179 | 0
  rSBA-MenW-135 [M 2], ≥1:128 |  | 90 | 178 |
  rSBA-MenY [M 0], ≥1:8: number analyzed (Participants) | 94 | 87 | 87 | 55
  rSBA-MenY [M 0], ≥1:8 | 57 | 53 | 53 | 30
  rSBA-MenY [M 1], ≥1:8: number analyzed (Participants) | 192 | 185 | 174 | 110
  rSBA-MenY [M 1], ≥1:8 | 192 | 180 | 103 | 71
  rSBA-MenY [M 2], ≥1:8: number analyzed (Participants) | 0 | 92 | 179 | 0
  rSBA-MenY [M 2], ≥1:8 |  | 91 | 178 |
  rSBA-MenY [M 0], ≥1:128: number analyzed (Participants) | 94 | 87 | 87 | 55
  rSBA-MenY [M 0], ≥1:128 | 38 | 37 | 34 | 20
  rSBA-MenY [M 1], ≥1:128: number analyzed (Participants) | 192 | 185 | 174 | 110
  rSBA-MenY [M 1], ≥1:128 | 192 | 178 | 79 | 38
  rSBA-MenY [M 2], ≥1:128: number analyzed (Participants) | 0 | 92 | 179 | 0
  rSBA-MenY [M 2], ≥1:128 |  | 91 | 178 |

6. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers
Description: The results were tabulated as geometric mean expressed in titers.
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 193 | 186 | 179 | 114
Titers
  rSBA-MenA [M 0]: number analyzed (Participants) | 84 | 77 | 72 | 46
  rSBA-MenA [M 0] | 15 [10 to 22.4] | 19 [12.2 to 29.5] | 24 [15 to 38.4] | 15.9 [9.2 to 27.5]
  rSBA-MenA [M 1]: number analyzed (Participants) | 193 | 183 | 163 | 100
  rSBA-MenA [M 1] | 3152.9 [2752.5 to 3611.4] | 3169.9 [2577.2 to 3898.8] | 24.2 [17.4 to 33.7] | 21.5 [14.5 to 32.1]
  rSBA-MenA [M 2]: number analyzed (Participants) | 0 | 90 | 178 | 0
  rSBA-MenA [M 2] |  | 2881.9 [2292 to 3623.6] | 1938.3 [1699.1 to 2211.2] |
  rSBA-MenC [M 0]: number analyzed (Participants) | 93 | 91 | 92 | 54
  rSBA-MenC [M 0] | 7.4 [5.7 to 9.6] | 9.1 [6.7 to 12.2] | 6.1 [4.9 to 7.7] | 7.6 [5.2 to 11.2]
  rSBA-MenC [M 1]: number analyzed (Participants) | 191 | 183 | 177 | 114
  rSBA-MenC [M 1] | 879.7 [763.1 to 1014] | 828.7 [672.4 to 1021.4] | 7.5 [6.1 to 9.3] | 691.4 [520.8 to 917.9]
  rSBA-MenC [M 2]: number analyzed (Participants) | 0 | 94 | 178 | 0
  rSBA-MenC [M 2] |  | 519.6 [391.7 to 689.2] | 386 [333.9 to 446.2] |
  rSBA-MenW-135 [M 0]: number analyzed (Participants) | 91 | 84 | 85 | 55
  rSBA-MenW-135 [M 0] | 19 [13.1 to 27.6] | 19.2 [13.3 to 27.7] | 24.8 [16.7 to 36.8] | 15.6 [9.8 to 25]
  rSBA-MenW-135 [M 1]: number analyzed (Participants) | 193 | 186 | 173 | 112
  rSBA-MenW-135 [M 1] | 4147 [3670.1 to 4685.8] | 4022.3 [3269.2 to 4948.8] | 25.2 [18.6 to 34.2] | 14.2 [10.2 to 19.7]
  rSBA-MenW-135 [M 2]: number analyzed (Participants) | 0 | 91 | 179 | 0
  rSBA-MenW-135 [M 2] |  | 3630.1 [2899.1 to 4545.4] | 2466.4 [2175.4 to 2796.4] |
  rSBA-MenY [M 0]: number analyzed (Participants) | 94 | 87 | 87 | 55
  rSBA-MenY [M 0] | 36.8 [24.7 to 54.8] | 45.4 [29.1 to 71] | 41.2 [26.7 to 63.4] | 32 [18.3 to 55.9]
  rSBA-MenY [M 1]: number analyzed (Participants) | 192 | 185 | 174 | 110
  rSBA-MenY [M 1] | 3461.8 [2990.1 to 4007.9] | 3167.7 [2521.9 to 3978.9] | 45.9 [33 to 63.9] | 47.2 [32.1 to 69.3]
  rSBA-MenY [M 2]: number analyzed (Participants) | 0 | 92 | 179 | 0
  rSBA-MenY [M 2] |  | 3010.4 [2325.3 to 3897.3] | 2446.9 [2088.5 to 2866.8] |

7. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off
Description: The cut-off for the assay were ≥ 0.3 microgram per milliliter (μg/mL) and ≥ 2.0 μg/mL, respectively.
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 51 | 47 | 47 | 29
Participants
  Anti-PSA [Month 0], ≥0.3: number analyzed (Participants) | 45 | 45 | 41 | 27
  Anti-PSA [Month 0], ≥0.3 | 4 | 1 | 1 | 1
  Anti-PSA [Month 1], ≥0.3: number analyzed (Participants) | 46 | 46 | 37 | 25
  Anti-PSA [Month 1], ≥0.3 | 46 | 45 | 1 | 1
  Anti-PSA [Month 2], ≥0.3: number analyzed (Participants) | 0 | 44 | 42 | 0
  Anti-PSA [Month 2], ≥0.3 |  | 44 | 42 |
  Anti-PSA [Month 0], ≥2.0: number analyzed (Participants) | 45 | 45 | 41 | 27
  Anti-PSA [Month 0], ≥2.0 | 0 | 0 | 0 | 0
  Anti-PSA [Month 1], ≥2.0: number analyzed (Participants) | 46 | 46 | 41 | 27
  Anti-PSA [Month 1], ≥2.0 | 46 | 44 | 1 | 0
  Anti-PSA [Month 2], ≥2.0: number analyzed (Participants) | 45 | 45 | 41 | 27
  Anti-PSA [Month 2], ≥2.0 | 0 | 43 | 40 | 0
  Anti-PSC [Month 0], ≥0.3: number analyzed (Participants) | 48 | 43 | 46 | 29
  Anti-PSC [Month 0], ≥0.3 | 1 | 1 | 2 | 0
  Anti-PSC [Month 1], ≥0.3: number analyzed (Participants) | 51 | 41 | 47 | 28
  Anti-PSC [Month 1], ≥0.3 | 51 | 41 | 2 | 28
  Anti-PSC [Month 2], ≥0.3: number analyzed (Participants) | 0 | 41 | 47 | 0
  Anti-PSC [Month 2], ≥0.3 |  | 41 | 47 |
  Anti-PSC [Month 0], ≥2.0: number analyzed (Participants) | 48 | 43 | 46 | 29
  Anti-PSC [Month 0], ≥2.0 | 1 | 0 | 0 | 0
  Anti-PSC [Month 1], ≥2.0: number analyzed (Participants) | 51 | 41 | 47 | 28
  Anti-PSC [Month 1], ≥2.0 | 50 | 41 | 0 | 26
  Anti-PSC [Month 2], ≥2.0: number analyzed (Participants) | 0 | 41 | 47 | 0
  Anti-PSC [Month 2], ≥2.0 |  | 41 | 43 |
  Anti-PSW-135 [Month 0], ≥0.3: number analyzed (Participants) | 44 | 43 | 40 | 26
  Anti-PSW-135 [Month 0], ≥0.3 | 1 | 1 | 2 | 0
  Anti-PSW-135 [Month 1], ≥0.3: number analyzed (Participants) | 44 | 47 | 41 | 26
  Anti-PSW-135 [Month 1], ≥0.3 | 44 | 43 | 2 | 0
  Anti-PSW-135 [Month 2], ≥0.3: number analyzed (Participants) | 0 | 44 | 41 | 0
  Anti-PSW-135 [Month 2], ≥0.3 | 0 | 43 | 41 | 0
  Anti-PSW-135 [Month 0], ≥2.0: number analyzed (Participants) | 44 | 43 | 40 | 26
  Anti-PSW-135 [Month 0], ≥2.0 | 0 | 0 | 1 | 0
  Anti-PSW-135 [Month 1], ≥2.0: number analyzed (Participants) | 44 | 47 | 41 | 26
  Anti-PSW-135 [Month 1], ≥2.0 | 40 | 39 | 2 | 0
  Anti-PSW-135 [Month 2], ≥2.0: number analyzed (Participants) | 0 | 41 | 41 | 0
  Anti-PSW-135 [Month 2], ≥2.0 |  | 36 | 29 |
  Anti-PSY [Month 0], ≥0.3: number analyzed (Participants) | 45 | 44 | 42 | 29
  Anti-PSY [Month 0], ≥0.3 | 1 | 1 | 0 | 0
  Anti-PSY [Month 1], ≥0.3: number analyzed (Participants) | 45 | 45 | 37 | 23
  Anti-PSY [Month 1], ≥0.3 | 45 | 43 | 1 | 0
  Anti-PSY [Month 2], ≥0.3: number analyzed (Participants) | 0 | 44 | 41 | 0
  Anti-PSY [Month 2], ≥0.3 |  | 44 | 41 |
  Anti-PSY [Month 0], ≥2.0: number analyzed (Participants) | 45 | 44 | 42 | 29
  Anti-PSY [Month 0], ≥2.0 | 0 | 0 | 0 | 0
  Anti-PSY [Month 1], ≥2.0: number analyzed (Participants) | 45 | 45 | 37 | 23
  Anti-PSY [Month 1], ≥2.0 | 40 | 42 | 1 | 0
  Anti-PSY [Month 2], ≥2.0: number analyzed (Participants) | 0 | 44 | 41 | 0
  Anti-PSY [Month 2], ≥2.0 |  | 40 | 34 |

8. Secondary Outcome: Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results for the assay were tabulated as geometric mean expressed in microgram per milliliter (μg/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 51 | 47 | 47 | 29
μg/mL
  Anti-PSA [M 0]: number analyzed (Participants) | 45 | 45 | 41 | 27
  Anti-PSA [M 0] | 0.17 [0.15 to 0.19] | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.18] | 0.16 [0.14 to 0.18]
  Anti-PSA [M 1]: number analyzed (Participants) | 46 | 46 | 37 | 25
  Anti-PSA [M 1] | 31.01 [23.73 to 40.52] | 33.15 [21.89 to 50.18] | 0.17 [0.13 to 0.22] | 0.16 [0.14 to 0.18]
  Anti-PSA [M 2]: number analyzed (Participants) | 0 | 44 | 42 | 0
  Anti-PSA [M 2] |  | 16.93 [12.39 to 23.13] | 12.28 [9.38 to 16.06] |
  Anti-PSC [M 0]: number analyzed (Participants) | 48 | 43 | 46 | 29
  Anti-PSC [M 0] | 0.16 [0.14 to 0.2] | 0.16 [0.14 to 0.17] | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.15]
  Anti-PSC [M 1]: number analyzed (Participants) | 51 | 41 | 47 | 28
  Anti-PSC [M 1] | 13.74 [10.68 to 17.67] | 23.52 [18.91 to 29.25] | 0.16 [0.15 to 0.17] | 7.99 [5.57 to 11.46]
  Anti-PSC [M 2]: number analyzed (Participants) | 0 | 41 | 47 | 0
  Anti-PSC [M 2] |  | 9.73 [7.82 to 12.12] | 5.84 [4.66 to 7.32] |
  Anti-PSW-135 [M 0]: number analyzed (Participants) | 44 | 43 | 40 | 26
  Anti-PSW-135 [M 0] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.16] | 0.17 [0.14 to 0.22] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 [M 1]: number analyzed (Participants) | 44 | 47 | 41 | 26
  Anti-PSW-135 [M 1] | 6.43 [4.92 to 8.4] | 4.15 [2.82 to 6.11] | 0.18 [0.14 to 0.22] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 [M 2]: number analyzed (Participants) | 0 | 44 | 41 | 0
  Anti-PSW-135 [M 2] |  | 3.99 [2.91 to 5.48] | 3.4 [2.52 to 4.59] |
  Anti-PSY [M 0]: number analyzed (Participants) | 45 | 44 | 42 | 29
  Anti-PSY [M 0] | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15]
  Anti-PSY [M 1]: number analyzed (Participants) | 45 | 45 | 37 | 23
  Anti-PSY [M 1] | 6.52 [4.91 to 8.65] | 9.42 [6.49 to 13.66] | 0.17 [0.13 to 0.21] | 0.15 [0.15 to 0.15]
  Anti-PSY [M 2]: number analyzed (Participants) | 0 | 44 | 41 | 0
  Anti-PSY [M 2] |  | 7.86 [6.04 to 10.23] | 4.76 [3.73 to 6.09] |

9. Secondary Outcome: Number of Seroprotected Subjects for Anti-tetanus Toxoid (Anti-TT)
Description: The cut-off for the assay was ≥ 0.1
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 186 | 180 | 176 | 110
Participants
  anti-TT [M 0], ≥0.1: number analyzed (Participants) | 186 | 177 | 171 | 108
  anti-TT [M 0], ≥0.1 | 177 | 161 | 155 | 99
  anti-TT [M 1], ≥0.1: number analyzed (Participants) | 184 | 180 | 174 | 110
  anti-TT [M 1], ≥0.1 | 184 | 177 | 173 | 99
  anti-TT [M 2], ≥0.1: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-TT [M 2], ≥0.1 |  | 177 | 176 |

10. Secondary Outcome: Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations
Description: The results for the assay were tabulated as geometric mean expressed in internationl units per milliliter (IU/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 186 | 180 | 176 | 110
IU/mL
  anti-TT [M 0]: number analyzed (Participants) | 186 | 177 | 171 | 108
  anti-TT [M 0] | 0.481 [0.417 to 0.554] | 0.39 [0.332 to 0.457] | 0.416 [0.354 to 0.489] | 0.393 [0.325 to 0.475]
  anti-TT [M 1]: number analyzed (Participants) | 184 | 180 | 174 | 110
  anti-TT [M 1] | 10.47 [9.131 to 12.007] | 7.941 [6.517 to 9.677] | 6.189 [5.404 to 7.089] | 0.374 [0.306 to 0.457]
  anti-TT [M 2]: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-TT [M 2] |  | 13.966 [12.199 to 15.987] | 8.236 [7.348 to 9.231] |

11. Secondary Outcome: Number of Subjects Seroprotected for Anti-diphtheria (Anti-D) ≥ the Cut-off
Description: The cut-off for the assay was ≥ 0.1
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 185 | 178 | 176 | 110
Participants
  anti-D [M 0], ≥0.1: number analyzed (Participants) | 185 | 174 | 170 | 106
  anti-D [M 0], ≥0.1 | 169 | 157 | 154 | 94
  anti-D [M 1], ≥0.1: number analyzed (Participants) | 184 | 178 | 174 | 110
  anti-D [M 1], ≥0.1 | 184 | 156 | 173 | 109
  anti-D [M 2], ≥0.1: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-D [M 2], ≥0.1 |  | 176 | 176 |

12. Secondary Outcome: Anti-diphtheria (Anti-D) Antibody Concentrations
Description: The results for the assay were tabulated as geometric mean expressed in internationl units per milliliter (IU/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 185 | 178 | 176 | 110
IU/mL
  anti-D [M 0]: number analyzed (Participants) | 185 | 174 | 170 | 106
  anti-D [M 0] | 0.477 [0.407 to 0.559] | 0.476 [0.397 to 0.57] | 0.437 [0.367 to 0.521] | 0.452 [0.355 to 0.574]
  anti-D [M 1]: number analyzed (Participants) | 184 | 178 | 174 | 110
  anti-D [M 1] | 7.636 [6.889 to 8.465] | 0.404 [0.335 to 0.487] | 7.292 [6.362 to 8.358] | 5.201 [4.243 to 6.376]
  anti-D [M 2]: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-D [M 2] |  | 8.561 [7.553 to 9.703] | 5.21 [4.623 to 5.872] |

13. Secondary Outcome: Number of Subjects Seroprotected for Anti-polio Type 1, 2 & 3 ≥ the Cut-off
Description: The cut-off for the assay was ≥ 1:8.
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 168 | 164 | 164 | 100
Participants
  anti-p1 [M 0]: number analyzed (Participants) | 168 | 161 | 156 | 100
  anti-p1 [M 0] | 158 | 143 | 142 | 90
  anti-p1 [M 1]: number analyzed (Participants) | 167 | 164 | 164 | 99
  anti-p1 [M 1] | 166 | 149 | 163 | 89
  anti-p1 [M 2]: number analyzed (Participants) | 0 | 160 | 162 | 0
  anti-p1 [M 2] |  | 159 | 161 |
  anti-p2 [M 0]: number analyzed (Participants) | 168 | 161 | 156 | 98
  anti-p2 [M 0] | 153 | 141 | 145 | 80
  anti-p2 [M 1]: number analyzed (Participants) | 167 | 164 | 163 | 98
  anti-p2 [M 1] | 166 | 147 | 161 | 80
  anti-p2 [M 2]: number analyzed (Participants) | 0 | 159 | 162 | 0
  anti-p2 [M 2] |  | 159 | 161 |
  anti-p3 [M 0]: number analyzed (Participants) | 168 | 161 | 157 | 100
  anti-p3 [M 0] | 155 | 148 | 143 | 88
  anti-p3 [M 1]: number analyzed (Participants) | 167 | 163 | 163 | 100
  anti-p3 [M 1] | 167 | 150 | 160 | 87
  anti-p3 [M 2]: number analyzed (Participants) | 0 | 160 | 161 | 0
  anti-p3 [M 2] |  | 159 | 159 |

14. Secondary Outcome: Anti-polio Type 1, 2 & 3 Titers
Description: The results for the assay were tabulated as geometric mean expressed in titers.
Time Frame: At month 0, 1 and 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 168 | 164 | 164 | 100
Titers
  anti-p1 [M 0]: number analyzed (Participants) | 168 | 161 | 156 | 100
  anti-p1 [M 0] | 84.2 [67.2 to 105.4] | 72.5 [55.6 to 94.5] | 83.6 [65.5 to 106.6] | 71.7 [51.7 to 99.6]
  anti-p1 [M 1]: number analyzed (Participants) | 167 | 164 | 164 | 99
  anti-p1 [M 1] | 984.4 [830.4 to 1167] | 74.2 [56.7 to 97.3] | 1308.5 [1073.2 to 1595.5] | 66.3 [46.6 to 94.4]
  anti-p1 [M 2]: number analyzed (Participants) | 0 | 160 | 162 | 0
  anti-p1 [M 2] |  | 1288.2 [1052.5 to 1576.6] | 1108.4 [913.5 to 1344.8] |
  anti-p2 [M 0]: number analyzed (Participants) | 168 | 161 | 156 | 98
  anti-p2 [M 0] | 76.8 [60.8 to 97] | 66.3 [50.9 to 86.5] | 65.6 [51.2 to 84.2] | 49.3 [34.9 to 69.6]
  anti-p2 [M 1]: number analyzed (Participants) | 167 | 164 | 163 | 98
  anti-p2 [M 1] | 1372 [1153.5 to 1631.9] | 70.3 [53.4 to 92.6] | 1540.4 [1253.2 to 1893.2] | 49.8 [34.5 to 71.9]
  anti-p2 [M 2]: number analyzed (Participants) | 0 | 159 | 162 | 0
  anti-p2 [M 2] |  | 1650.5 [1358.5 to 2005.3] | 1174.5 [961.4 to 1434.8] |
  anti-p3 [M 0]: number analyzed (Participants) | 168 | 161 | 157 | 100
  anti-p3 [M 0] | 104.4 [81.1 to 134.4] | 99.8 [77.5 to 128.5] | 113.2 [86.9 to 147.5] | 102.9 [72.8 to 145.4]
  anti-p3 [M 1]: number analyzed (Participants) | 167 | 163 | 163 | 100
  anti-p3 [M 1] | 2295.6 [1952.1 to 2699.4] | 96.6 [74.2 to 125.8] | 2034.3 [1594.9 to 2594.8] | 85.3 [58.7 to 124.1]
  anti-p3 [M 2]: number analyzed (Participants) | 0 | 160 | 161 | 0
  anti-p3 [M 2] |  | 2478 [2049.2 to 2996.4] | 1655.1 [1308.9 to 2092.9] |

15. Secondary Outcome: Numbers of Seroprotected Subjects for Anti-PRP ≥ the Cut-off
Description: The cut-off for the assay was ≥ 1.0
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 185 | 179 | 176 | 110
Participants
  anti-PRP [M 0] ≥1.0: number analyzed (Participants) | 185 | 175 | 171 | 108
  anti-PRP [M 0] ≥1.0 | 73 | 64 | 65 | 34
  anti-PRP [M 1] ≥1.0: number analyzed (Participants) | 184 | 179 | 173 | 110
  anti-PRP [M 1] ≥1.0 | 183 | 70 | 170 | 34
  anti-PRP [M 2] ≥1.0: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-PRP [M 2] ≥1.0 |  | 172 | 170 |

16. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: The results for the assay were tabulated as geometric mean expressed in microgram per milliliter (μg/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 185 | 179 | 176 | 110
μg/mL
  anti-PRP [M 0]: number analyzed (Participants) | 185 | 175 | 171 | 108
  anti-PRP [M 0] | 0.806 [0.658 to 0.987] | 0.665 [0.528 to 0.839] | 0.766 [0.596 to 0.986] | 0.585 [0.449 to 0.762]
  anti-PRP [M 1]: number analyzed (Participants) | 184 | 179 | 173 | 110
  anti-PRP [M 1] | 25.556 [21.358 to 30.579] | 0.711 [0.56 to 0.904] | 31.165 [25.142 to 38.631] | 0.55 [0.42 to 0.72]
  anti-PRP [M 2]: number analyzed (Participants) | 0 | 177 | 176 | 0
  anti-PRP [M 2] |  | 12.239 [10.392 to 14.414] | 21.023 [17.036 to 25.942] |

17. Secondary Outcome: Number of Seroprotected Subjects for Anti-HBs ≥ the Cut-offs
Description: The cut-offs for the assay were ≥ 10 mIU/mL and ≥ 100 mIU/mL respectively .
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 181 | 174 | 169 | 106
Participants
  anti-HBS [M 0] ≥10: number analyzed (Participants) | 180 | 169 | 166 | 102
  anti-HBS [M 0] ≥10 | 173 | 158 | 155 | 95
  anti-HBS [M 1] ≥10 | 180 | 160 | 166 | 100
  anti-HBS [M 2] ≥10: number analyzed (Participants) | 0 | 173 | 168 | 0
  anti-HBS [M 2] ≥10 |  | 172 | 167 |
  anti-HBS [M 0] ≥100: number analyzed (Participants) | 180 | 169 | 166 | 102
  anti-HBS [M 0] ≥100 | 92 | 80 | 75 | 46
  anti-HBS [M 1] ≥100 | 169 | 85 | 155 | 46
  anti-HBS [M 2] ≥100: number analyzed (Participants) | 0 | 173 | 168 | 0
  anti-HBS [M 2] ≥100 |  | 168 | 158 |

18. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: The results for the assay were tabulated as geometric mean expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 181 | 174 | 169 | 106
mIU/mL
  anti-HBS [M 0]: number analyzed (Participants) | 180 | 169 | 166 | 102
  anti-HBS [M 0] | 111.6 [90.9 to 136.9] | 92.8 [75.3 to 114.4] | 101.2 [81.5 to 125.7] | 85.6 [65.7 to 111.5]
  anti-HBS [M 1] | 2048.4 [1589.3 to 2640] | 95 [74.8 to 120.6] | 1711.6 [1292.7 to 2266.3] | 101.6 [75.5 to 136.7]
  anti-HBS [M 2]: number analyzed (Participants) | 0 | 173 | 168 | 0
  anti-HBS [M 2] |  | 2392.3 [1841.7 to 3107.4] | 1241 [976.2 to 1577.7] |

19. Secondary Outcome: Number of Subjects With a Vaccine Response to PT, FHA and PRN Antigens
Description: Vaccine response to these antigens is defined as appearance of antibodies in subjects who were seronegative (antibody concentration < 5 EL.U/mL) at pre-vaccination or as at least a 2-fold increase in post-over pre-vaccination antibody concentrations in subjects seropositive at pre-vaccination.
  The analysis was based only on subjects receiving experimental vaccination.
Time Frame: 1 month after vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component prior to (M0) and after vaccination (M1).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group
Number analyzed (Participants) | 190 | 178 | 174
Participants
  Anti-PT: number analyzed (Participants) | 190 | 176 | 173
  Anti-PT | 180 | 169 | 163
  Anti-FHA: number analyzed (Participants) | 190 | 173 | 172
  Anti-FHA | 184 | 159 | 158
  Anti-PRN | 186 | 173 | 172

20. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: The results were tabulated as geometric mean expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At month 0, month 1 and month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 194 | 188 | 182 | 114
EL.U/mL
  Anti-PT [M 0]: number analyzed (Participants) | 193 | 187 | 182 | 112
  Anti-PT [M 0] | 11 [10 to 12] | 10 [8 to 11] | 10 [9 to 12] | 11 [9 to 13]
  Anti-PT [M 1]: number analyzed (Participants) | 191 | 180 | 178 | 109
  Anti-PT [M 1] | 86 [77 to 95] | 8 [7 to 9] | 85 [75 to 96] | 9 [7 to 10]
  Anti-PT [M 2]: number analyzed (Participants) | 0 | 177 | 179 | 0
  Anti-PT [M 2] |  | 91 [80 to 102] | 63 [55 to 71] |
  Anti-FHA [M 0]: number analyzed (Participants) | 193 | 183 | 181 | 111
  Anti-FHA [M 0] | 51 [44 to 59] | 55 [46 to 66] | 49 [41 to 57] | 55 [44 to 68]
  Anti-FHA [M 1]: number analyzed (Participants) | 191 | 183 | 178 | 110
  Anti-FHA [M 1] | 542 [492 to 597] | 48 [40 to 58] | 544 [485 to 611] | 55 [42 to 71]
  Anti-FHA [M 2]: number analyzed (Participants) | 0 | 178 | 176 | 0
  Anti-FHA [M 2] |  | 664 [664 to 750] | 413 [366 to 465] |
  Anti-PRN [M 0] | 26 [23 to 31] | 26 [22 to 31] | 21 [17 to 24] | 23 [18 to 28]
  Anti-PRN [M 1]: number analyzed (Participants) | 190 | 184 | 179 | 112
  Anti-PRN [M 1] | 470 [411 to 537] | 23 [19 to 27] | 450 [387 to 522] | 21 [16 to 26]
  Anti-PRN [M 2]: number analyzed (Participants) | 0 | 178 | 178 | 0
  Anti-PRN [M 2] |  | 583 [502 to 676] | 336 [286 to 395] |

21. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms Post-meningococcal Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any local symptom irrespective of intensity grade. Grade 3 Pain was defined as crying when limb was moved/ spontaneously painful.
Time Frame: During the 4-day (Days 0-3) follow-up period after Nimenrix or Meningitec vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects with the symptom sheet filled-in after meningococcal vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 220 | 217 | 219 | 126
Participants
  Any Pain | 49 | 30 | 35 | 16
  Grade 3 Pain | 3 | 0 | 1 | 1
  Any Redness | 70 | 74 | 56 | 36
  Grade 3 Redness | 3 | 8 | 8 | 2
  Any Swelling | 42 | 36 | 36 | 23
  Grade 3 Swelling | 2 | 3 | 7 | 0

22. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms Post-combined Diphtheria Vaccination
Description: The analysis was based only on subjects receiving combined-diphtheria vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after Infanrix-hexa vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects with the symptom sheet filled-in after the Infanrix-hexa vaccination. Subjects in the Meningitec Group did not receive any Infanrix-hexa and hence are not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group
Number analyzed (Participants) | 220 | 209 | 221
Participants
  Any Pain | 60 | 65 | 64
  Grade 3 Pain | 6 | 5 | 10
  Any Redness | 70 | 77 | 99
  Grade 3 Redness | 11 | 14 | 27
  Any Swelling | 48 | 53 | 74
  Grade 3 Swelling | 12 | 14 | 22

23. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms Following Each Dose
Description: Solicited general symptoms assessed were drowsiness, fever, irritability and loss of appetite. Any was defined as occurrence of any general symptom irrespective of intensity grade and relationship.
  Subjects in the Nimenrix + Infanrix-hexa Group did not receive a second dose of vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination dose 1 (D1) and second dose (D2)
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 220 | 218 | 221 | 126
Participants
  Drowsiness, D1 | 85 | 56 | 80 | 29
  Fever, D1 | 80 | 41 | 71 | 15
  Irritability, D1 | 83 | 63 | 75 | 25
  Loss of appetite, D1 | 51 | 46 | 51 | 15
  Drowsiness, D2 | 0 | 63 | 56 | 0
  Fever, D2 | 0 | 60 | 37 | 0
  Irritability, D2 | 0 | 75 | 50 | 0
  Loss of appetite, D2 | 0 | 54 | 38 | 0

24. Secondary Outcome: Number of Subjects Reporting Any Rash
Description: Any was defined as occurrence of at least one symptom experienced.
Time Frame: Day 0 - Month 7
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 222 | 220 | 224 | 127
Participants | 13 | 25 | 22 | 12

25. Secondary Outcome: Number of Subjects Reporting Any New Onset of Chronic Illnesses (NOCIs)
Description: Any was defined as occurrence of at least one symptom experienced.
Time Frame: Day 0 - Month 7
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 222 | 220 | 224 | 127
Participants | 1 | 2 | 6 | 1

26. Secondary Outcome: Number of Subjects Reporting Any Conditions Prompting Emergency Room Visits (ER)
Description: Any was defined as occurrence of at least one symptom experienced.
Time Frame: Day 0 - Month 7
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 222 | 220 | 224 | 127
Participants | 5 | 3 | 14 | 6

27. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs) After the First Dose
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined as an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Occurring within Day 0-30 following vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 222 | 220 | 224 | 127
Participants | 71 | 81 | 83 | 42

28. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs) After the Second Dose
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined as an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
  The analysis was based only on subjects receiving a second dose of vaccination.
Time Frame: Occurring within Day 0-30 following vaccination
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Infanrix-Hexa Group
Number analyzed (Participants) | 215 | 221
Participants | 87 | 79

29. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: From dose 1 (Month 0) up to study end (Month 7)
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
Number analyzed (Participants) | 222 | 220 | 224 | 127
Participants | 10 | 8 | 11 | 6

ADVERSE EVENTS:
Time Frame: SAEs were reported throughout the entire study period (Day 0 - Month 7). Solicited symptoms were reported during a 4-day period (Day 0-Day 3) after any vaccine dose, while unsolicited AEs were collected within 31 days (Days 0-30) after vaccination.
Description: The solicited local and general symptoms were only collected for those subjects who filled-in their symptom sheets.
Arm/Group | Nimenrix + Infanrix-hexa Group | Nimenrix Group | Infanrix-Hexa Group | Meningitec Group
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/220 | 1/224 | 0/127
Serious Adverse Events (participants affected / at risk) | 10/222 | 8/220 | 11/224 | 6/127
Other Adverse Events (participants affected / at risk) | 166/222 | 183/220 | 185/224 | 75/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix + Infanrix-hexa Group (N=222) | Nimenrix Group (N=220) | Infanrix-Hexa Group (N=224) | Meningitec Group (N=127)
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile convulsion (Nervous system disorders) | 2 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0
Drowning (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Coxsackie viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix + Infanrix-hexa Group (N=222) | Nimenrix Group (N=220) | Infanrix-Hexa Group (N=224) | Meningitec Group (N=127)
Bronchitis (Infections and infestations) | 7 (7) | 16 (18) | 12 (13) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (11) | 5 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 51 (51) | 78 (100) | 68 (89) | 15 (15)
Erythema (Skin and subcutaneous tissue disorders) | 91 (91) | 102 (151) | 103 (155) | 36 (37)
Gastroenteritis (Infections and infestations) | 6 (6) | 18 (20) | 18 (18) | 4 (4)
Irritability (Psychiatric disorders) | 83 (83) | 100 (139) | 93 (125) | 25 (25)
Nasopharyngitis (Infections and infestations) | 3 (3) | 12 (15) | 11 (12) | 2 (2)
Otitis media (Infections and infestations) | 4 (4) | 11 (12) | 7 (7) | 5 (5)
Pain (General disorders) | 68 (69) | 75 (95) | 69 (99) | 16 (16)
Pyrexia (General disorders) | 83 (86) | 90 (114) | 89 (114) | 17 (17)
Rhinitis (Infections and infestations) | 9 (11) | 16 (17) | 10 (10) | 1 (1)
Somnolence (Nervous system disorders) | 85 (85) | 89 (119) | 95 (136) | 29 (29)
Swelling (General disorders) | 64 (64) | 66 (89) | 85 (110) | 23 (23)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 27 (30) | 24 (27) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.